CLINICAL TRIAL: NCT06498544
Title: HighCycle Study: Effect of High Altitude on Sleep Disordered Breathing in Women Related to Their Menstrual Cycle Phase. A Prospective Cohort Study at 3600 m.
Brief Title: HighCycle Study: Effect of High Altitude on Sleep Disordered Breathing in Women Related to Their Menstrual Cycle Phase
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government); University Hospital Heidelberg (Other); Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Other Study IDs: HighCycle_SDB_MCP
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Sleep-Disordered Breathing
Keywords: Periodic breathing; Hypoxia; Prevention; Acetazolamide; Women; Altitude
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women in luteal MCP: Women being in their luteal MCP on the day of ascent to high altitude.
  Interventions: Other: Exposure to 3600 m
- Women in follicular MCP: Women being in their follicular MCP on the day of ascent to high altitude.
  Interventions: Other: Exposure to 3600 m

INTERVENTIONS:
Other: Exposure to 3600 m — Participants will travel to and stay for 2 nights at an altitude of 3600 m.

SUMMARY:
Prospective cohort study investigating the menstrual cycle phase (MCP) dependent sleep disordered breathing (SDB) in women travelling to 3600 m.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Healthy, non-smoking women, age 18-44 years, without any diseases and need of regular medication (including oral contraceptives).
* BMI >18 kg/m2 and <30 kg/m2
* Born, raised and currently living at altitudes <1000 m
* Written informed consent
* Premenopausal, eumenorrheic cycle

Exclusion Criteria:

* Other types of contraceptives (hormonal intrauterine device, vaginal ring, subcutaneous injections or implants, among others)
* Pregnancy or nursing
* Anaemic (haemoglobin concentration <10g/dl)
* Any altitude trip <4 weks before the study
* Allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, non-smoking, premenopausal women, age 18-44 years, without any disease and need of regular medication (including oral contraceptives).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Nocturnal oxygen saturation (SpO2) | Night 1 at 760 m and Night 1 at 3600 m
  MCP-related difference in altitude-induced change in the mean nocturnal oxygen saturation measured by pulse oximetry.

SECONDARY OUTCOMES:
Nocturnal oxygen desaturation index (ODI) | Night 1 at 760 m and Night 1 at 3600 m
  MCP-related difference in altitude-induced change in the ODI (number of ∆SpO2 >3% per hour time in bed measured by pulse oximetry).
Nocturnal oxygen desaturation index (ODI) | Night 1 at 760 m and Night 2 at 3600 m
  MCP-related difference in altitude-induced change in the ODI (number of ∆SpO2 >3% per hour time in bed measured by pulse oximetry).
Apnea/hypopnea index (AHI) | Night 1 at 760 m and Night 1 at 3600 m
  MCP-related difference in altitude-induced change in the mean number of apneas/hypopneas per hour.
Apnea/hypopnea index (AHI) | Night 1 at 760 m and Night 2 at 3600 m
  MCP-related difference in altitude-induced change in the mean number of apneas/hypopneas per hour.
Subjective sleep quality | Night 1 at 760 m and Night 1 at 3600 m
  MCP-related difference in altitude-induced change in subjective sleep quality assessed by a 100-mm visual analog scale.
Subjective sleep quality | Night 1 at 760 m and Night 2 at 3600 m
  MCP-related difference in altitude-induced change in subjective sleep quality assessed by a 100-mm visual analog scale.
Nocturnal oxygen saturation (SpO2) | Night 1 at 760 m and Night 2 at 3600 m
  MCP-related difference in altitude-induced change in the mean nocturnal oxygen saturation measured by pulse oximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Furian, Prof. Dr., Study Chair — University of Zurich; Talant Sooronbaev, Prof. Dr., Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Gorod Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided